CLINICAL TRIAL: NCT03603613
Title: Youth Functioning and Organizational Success for West African Regional Development: Pilot
Brief Title: Youth FORWARD Phase 1 YRI and EPP Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: German Society for International Cooperation (Other); Caritas Freetown (Other); University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.068.01
Record Dates: First submitted 2018-05-18; First posted 2018-07-27 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Mental Health Disorder; Mental Health Impairment; Psychosocial Impairment; Emotional Dysfunction
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: A cluster randomized three-arm trial will be employed in the pilot phase in the same districts as the scale-up study. Youth (N=180, 18-26 years old, 50% female), stratified by gender, will be randomized into the three study arms. Once youth are enrolled into the study, they will be assigned to community level sites based on geographical location. Each of these community level sites will make up one cluster. The clusters will then be randomly assigned into the three study arms so that sixty youth will be randomized into the youth employment promotion program (EPP) arm, sixty youth will be randomized into the YRI+EPP arm, and sixty youth will be randomized into the control arm . The pilot study will last approximately 12 weeks and data will be collected at baseline and post-intervention. Further, we will survey 120 third-party reporters for a total pilot study sample size of 300 participants.
Who Masked: Outcomes Assessor
Masking Description: Under the supervision of Innovations for Poverty Action (IPA) Sierra Leone, local research assistants (blind to site and youth condition assignments) will conduct all screening, baseline, and follow up quantitative assessments. Ongoing data collection at all sites will include youth attendance and satisfaction with YRI content, counselor satisfaction with content and delivery via scales and qualitative exit interviews, as well as monitored audio-recording of all sessions for fidelity by an independent expert rater hired by CARITAS. The expert fidelity monitor will be a skilled YRI trainer and supervisor from our prior RCT and will not be a part of the standard CTS training condition nor the ICT Seed Team, thus allowing them to provide impartial and blinded fidelity ratings of all audio-transcripts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPP: Entrepreneurship Programme (Experimental): EPP: Entrepreneurship Programme: Youth randomized into the EPP-only arm will receive GIZ's employment programming within two weeks after the completion of the baseline assessments. The GIZ-supported EPP program includes six training modules. The modules include skills related to entrepreneurship, financial literacy, and skills building.
  Interventions: Behavioral: EPP
- EPP+YRI (Experimental): EPP+YRI: Youth randomized into the EPP+YRI arm will begin the Entrepreneurship programme within two weeks of baseline assessments. The entrepreneurship modules will occur for 15 days for 5 hours each day, 5 days per week. Immediately following the EPP, youth will begin receiving the YRI. The YRI curriculum (12 modules), will be delivered twice weekly over the course of 6 weeks. Each session lasts approximately 90-minutes, with additional time taken as needed. These sessions assume a peer-to-peer group learning format deemed culturally appropriate for a setting like Sierra Leone where limited resources for mental health services exist. Once youth complete the YRI they will complete a post-intervention quantitative assessment.
  Interventions: Behavioral: YRI; Behavioral: EPP
- Control (No Intervention): Control: Youth randomized into the control arm will be quantitatively assessed at the same time points as youth randomized into the two treatment arms (baseline and post-intervention). Due to access to funding and feasibility, youth in the control arm will not have the opportunity to receive the YRI once the study period concludes. However, GIZ is conducting a phased roll out of their EPP programming, meaning they will offer their EPP throughout 2018 past their participation in Youth FORWARD. The list of youth from the control group will be provided to GIZ so they can participate in the future phases. Youth will also be compensated for their participation in our quantitative assessments.

INTERVENTIONS:
Behavioral: YRI — The YRI is designed to assist youth facing complex problems using evidence-based treatments that have been tested and shown to work well in other settings and cultures. The YRI has three specific goals: 1) develop emotion regulation skills for healthy coping; 2) develop problem-solving skills to assist with achieving goals, and; 3) improve interpersonal skills to enable healthy relationships and effective communication. It integrates six CBT-based, empirically-supported practice elements shown to have transdiagnostic efficacy across disorders ranging from major depressive disorder to PTSD and conduct disorders. The YRI's six evidence-based components are delivered in three phases common in trauma-informed interventions: stabilization, integration, and connection.
  Other Names: Youth Readiness Intervention
  Arms: EPP+YRI
Behavioral: EPP — The youth capacity development component of GIZ's EPP includes the following core components: financial literacy, entrepreneurship, and vocational training delivered through six modules (agro-processing, solar photovoltaic installation and maintenance, governance and conflict resolution, psychosocial competencies, entrepreneurship, employability). Youth will be trained at training sites and have access to a youth center in the area. These centers will have agricultural equipment and machinery available for youth to use. Our YRI curriculum will be used for the psychosocial competency training module.
  Other Names: Youth Employment Promotion Programme
  Arms: EPP+YRI; EPP: Entrepreneurship Programme

SUMMARY:
Objectives: The objectives of this research proposal are to study the delivery of an evidence-based mental health intervention in the alternate setting of youth employment programs tied to regional economic development and to examine the use of an Interagency Collaborative Team Approach (ICTA) as an implementation scale-up strategy that addresses the human resource shortage and related access to care and capacity challenges in low- and middle-income countries (LMICs). Specifically, this study aims to examine the incorporation of the evidence-based Youth Readiness Intervention (YRI) into a program that promotes employment among youth through a pilot study and scale-up intervention study in Sierra Leone.

Study population: The study population includes youth participants, ages 18-26, with elevated t-scores on assessments of functional impairment and emotional dysregulation, who live in the Kailhun District of Sierra Leone.

Pilot study design: A cluster randomized three-arm trial will be employed in the pilot phase in the same districts as the scale-up study. Youth participants (N=180, 18-26 years old, 50% female), stratified by gender, will be randomized into the three study arms. Once youth participants are enrolled into the study, they will be assigned to community level sites based on geographical location. Each of these community level sites will make up one cluster. The clusters will then be randomly assigned into the three study arms so that sixty youth participants will be randomized into the youth entrepreneurship training (EPP) arm, sixty youth participants will be randomized into the YRI+EPP arm, and sixty youth participants will be randomized into the control arm . The pilot study will last approximately 12 weeks and data will be collected at baseline and post-intervention. Further, investigators will survey 120 third-party reporters for a total pilot study sample size of 300 participants.

Pilot study primary outcomes: The primary outcomes of the pilot study are to assess implementation science aspects related to a new partnership with the Deutsche Gesellschaft für Internationale Zusammenarbeit's (GIZ), who will fund and deliver the entrepreneurship training. This will include pretesting the measures battery, assessing the logistics of integrating the YRI into the entrepreneurship training, and testing use of the Interagency Collaborative Team Approach to training, supervision, and fidelity monitoring.

DETAILED DESCRIPTION:
Pilot study aims

1. To examine the psychometric properties of an existing measures battery as well as a new battery for third-party reporting,
2. To assess and adjust as needed structures for training and supervision, including the ICTA, and methods for conducting process evaluations of implementation procedures, and;
3. To assess the feasibility of integrating the YRI into the entrepreneurship training (EPP) and using the ICTA to deliver an evidence-informed intervention in Sierra Leone.

Study design

The investigators are proposing to conduct a small cluster randomized pilot study with a sample of 180 youth participants, aged 18 to 26 years old. Gender within the sample will be evenly split with 50% male and 50% female youth participants. GIZ will initiate recruitment of and selection of youth participants. An electronic database will only be used by members of the research team to contact the youth participants about participating in the research study. An additional screening will be completed to ensure candidates meet specific study eligibility criteria. Given the socioemotional aims of the YRI, youth participants must demonstrate impaired functioning and emotional dysregulation.

The research team will use the information in the database to contact the EPP-selected individuals about participating in our study. Research team members will first attempt to reach EPP-selected individuals by telephone, using the telephone numbers provided in the database. If an EPP-selected individual is not reachable by telephone, the research team will attempt to locate the youth participants at their residence, using the information in the database. Because GIZ is a well-known organization in Sierra Leone that has been working in the country for many decades and supports a number of employment programs in Kono, Kailahun and Koinadugu districts, the investigators do not expect this method of contacting youth to cause them any adverse effects.

During the in-person appointment, the research team member will go through the informed consent process for the screening, the potential participant will give consent (or not) and the research team member will conduct the mental health screening. After this process, these potential participants will be told to wait for follow-up communication from the research team. Study investigators have used similar procedures in past studies with success when contacting potential study participants.

After all candidates have been screened, a list of those who meet study criteria will be created and youth will be assigned to community level sites based on geographical location. Each of these community level sites will make up one cluster. The clusters will be randomized into three arms - sixty youth participants will be randomized to receive the EPP only, sixty youth participants will be randomized to receive YRI+EPP, and sixty youth participants will be randomized into the control group. At least 180 youth participants will be recruited assuming 15-20% attrition of subjects, informed by previous work in the region. Given gender and cultural norms in Sierra Leone, the YRI+EPP groups will be segregated by sex and these groups will be led by same-sex facilitators.

The pilot will be conducted in Kailhun District, which is one of the districts where GIZ operates their employment program. This is also a districts where GIZ has historically worked.

Once the SPs have been on boarded, the in-country leadership team will meet with SP staff to discuss the YRI and EPP in-depth and assess interest in being a part of the seed team. Selection of the seed team will be followed by a two-week training, which includes the YRI and ICTA.

Although this pilot involves a small sample size and is only powered to detect large differences between the intervention groups (YRI+EPP and EPP-only) and control group (no treatment), investigators are most interested in assessing the feasibility of integrating the YRI into the EPP and using the ICTA to deliver an evidence-informed intervention in a setting like Sierra Leone while maintaining intervention quality and improving delivery, as well as pretesting the measures battery before the tools are used in the full scale-up study. The proposed pilot study design will allow study investigators to examine the psychometric properties of measures and do a preliminary assessment on feasibility of program integration and seed team functioning and general patterns of improvement whereby investigators expect to see greater improvement among youth in the YRI+EPP compared to EPP only.

Intervention delivery

Both the YRI and EPP will be delivered over three months. The YRI, which typically assumes a three-month delivery period (12 sessions in total, 1 delivered per week), will be delivered with two sessions per week allowing for a 1.5-month delivery period during the pilot phase. Youth participants will then complete the business skills modules of the EPP, which are expected to take another 1.5 months. While the scale-up study allows for the YRI to be delivered (0-3 months) followed by the EPP (3-6 months), the pilot approach will condense the implementation of the YRI to provide sufficient time to initiate pilot-driven changes and obtain Institutional Review Board (IRB) and local approvals before the scale-up is launched.

YRI facilitators will be selected from staff at the SPs selected by GIZ to deliver the EPP training modules. Training and utilization of staff within the ICTA model addresses core issues of sustainability within the pilot and larger scale-up study. The in-country leadership team will assess agency staff to determine those best suited to deliver the YRI+EPP, especially as it concerns this innovative approach to supervision and service delivery.

A sample of YRI facilitators will be selected to form a seed team as part of the ICTA within this pilot study. The seed team will work across study sites to engage in routine information sharing to promote ongoing intervention fidelity and promote cross-site learning. Those chosen to be a part of the seed team will receive training on this approach by in-country experts (Dr. Akinsulure-Smith and trained Caritas Freetown research team members) who have experience with previous YRI research in Sierra Leone. By incorporating the ICTA into the pilot, study investigators will be able to utilize the pilot seed team to train and supervise the larger team for the scale-up study.

Monitoring and evaluation

Data will be collected pre- and post-intervention by a strong team of in-country experts. Innovations for Poverty Action (IPA) will oversee and conduct quantitative data collection (youth assessment battery, seed team assessment battery, dissemination and implementation measures) and analysis while Caritas Freetown will oversee and conduct qualitative data collection as well as the assessment battery for the third-party reporters. IPA is a lead institution for designing randomized control and randomized cluster applied research on economic and health outcomes in a number of LMICs and has worked with Dr. Betancourt in varying capacities in Sierra Leone.

From previous iterations of the YRI in Sierra Leone, the quantitative assessment battery for youth participants underwent a thorough development, translation and validation process. All survey tools were subjected to forward and backward translation from English to Sierra Leonean Krio utilizing the WHO process of translation and adaptation of instruments, Measures have been subjected to cognitive testing to ensure comprehension and cultural relevance in assessing mental health, daily functioning, and other life outcomes. However, measures on socioeconomic status and economic self-sufficiency did not perform well in the GCC pilot study. Study investigators have explored the reasons why and revised the tool used and selected new measures, both of which will need to be piloted before being broadly used in the scale-up study. Since the impact of the YRI on socioeconomic status and economic self-sufficiency of youth participants is one of the aspects of the scale-up study investigators will be assessing, it is vital to test these new measures to get a sense of appropriateness and performance before including them in the scale-up study. The measures utilized in the pilot study will be refined and utilized in the scale-up. IPA frequently hires local individuals for short-term data collection assignments. To develop skills and capacity and promote consistency, IPA makes an effort to hire the same individuals whenever data collection opportunities arise. Thus, over time, these individuals have gained experience in data collection and data management and have been trained in all aspects of the research process by IPA permanent, experienced, qualified staff. IPA maintains a database of these individuals, and this will be used to select the data collection team who will work on our pilot and scale-up studies.

ELIGIBILITY:
Inclusion Criteria: Youth aged 18-26 will be included in the Youth FORWARD scale-up study based upon eligibility to the employment program, focusing specifically on socioeconomic status and willingness and interest in participation in an employment program, as well as mental health screening, which will include questions on daily functioning and emotional regulation.

Specifically, inclusion criteria for the youth sample is:

* be Sierra Leonean,
* be female or male aged 18-26,
* be considered a vulnerable youth who is disengaged from both education and employment programs,
* have elevated t-scores on functional impairment based on thresholds from our previous research using questions adapted from the World Health Organization Disability Assessment Schedule (WHODAS)54 and,
* have elevated t-scores (62.5 or above) on the Disturbances in Emotion Regulation Scale (DERS).55

Inclusion criteria for agencies in this study is:

* be a "service provision agency" in Sierra Leone,
* have a minimum of two experts employed, one with subject-specific knowledge and; experience, and another with pedagogical experience in adult education and working with youth with low literacy, and
* sign a Memorandum Of Understanding (MOU) with Boston College (BC) regarding intellectual property of the YRI.

Inclusion criteria for facilitators in this study is:

* be employed by one of the agencies selected in GIZ's competitive bidding process, and
* agree to participation in the ICTA which utilizes an enhanced supervision structure throughout the intervention.

Inclusion criteria for third-party reporters in this study is:

* be over age 18,
* be nominated by the youth participant,
* provide oral consent to participate in the quantitative assessments, and
* have daily to weekly contact with the youth participant throughout the duration of this scale-up study, which will be assess via verbal confirmation when obtaining oral consent.

Inclusion criteria for agency leaders is:

* must be a part of one of the agencies selected in GIZ's competitive bidding process and,
* must hold a leadership position in the agency.

Exclusion Criteria:

Exclusion criteria for the youth:

Youth will be excluded from the study if they do not fulfill the inclusion criteria or present with: -severe mental illness (e.g., psychosis), or

-developmental disability that precludes comprehension of the intervention content and assessments (as determined by a study social worker using the World Health Organization Disability Assessment Screener within the Youth Screening Tool available in Appendix C).

Specifically, mental health exclusion criteria are:

* severe, active suicidality or psychosis as assessed via the MINI-KID diagnostic assessment administered by a study social worker and,
* serious cognitive impairments that might preclude one's ability to comprehend informed consent and complete study assessments as determined by a study social worker, as assessed via the Youth Screening tool (Appendix C).

Youth who report active suicidality or symptoms of psychosis requiring more intensive mental health care will be referred for immediate individual mental health services

Exclusion criteria for the agencies:

Agencies will be excluded from participation if:

* they are not considered a "service provision agency", and
* if they do not have a minimum of two experts employed (one with subject-specific knowledge and experience, and another with pedagogical experience in adult education and working with youth with low literacy)

Those holding leadership positions within the agencies selected to deliver the intervention will be excluded from participation in the qualitative interviews if:

* they are not employed at the agencies selected, or
* are not considered to be in a leadership position within the agency.

Exclusion criteria for the facilitators:

Facilitators will be excluded from participation in delivering the intervention if:

* they are unable to deliver core components of the YRI and EPP intervention, and
* if they are unable to meet the logistical demands of the ICTA.

Exclusion criteria for the third-party reporters:

The third-party reporter will be excluded from the study if:

* they are under age 18
* present with severe mental illness (e.g., psychosis), or
* developmental disability that precludes comprehension of the intervention content and assessments (as determined by a study social worker), and
* does not have at least monthly contact with the youth participant

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 297 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Youth-level outcome measures: emotion regulation | baseline and 3-months (post-intervention)
  Change in youth mental emotion regulation will be assessed via the following measure:
  • Difficulties in Emotion Regulation (DERS), clinical threshold for emotion dysregulation set at a score of 62.5, range of scores is from 36-180, higher scores denote higher levels of emotion dysregulation

SECONDARY OUTCOMES:
Youth-level outcome measure: youth employment and economic self-sufficiency | baseline and 3-months (post-intervention)
  Change regarding youth employment and economic self-sufficiency will be assessed via a self-developed Income Generating Activities and Well-being Measure. This measures produces indicators, there are no scores that we pull from this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, Sc.D., M.A., Principal Investigator — Boston College
Locations (1):
- CARITAS, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: No
All hard copies of data will be stored in locked cabinets to which only the local PIs, study managers, and research assistants have access. After completion of an assessment with a study participant, data with study ID numbers will be placed in a subject binder in a separate locked file cabinet while waiting for data entry. Once data is entered into computer files and password protected, only the local PIs, study managers, and research assistants will have access to these files. The Boston-based research team will only have access to de-identified data.

REFERENCES:
- [Derived] Bond L, Farrar J, Borg RC, Keegan K, Journeay K, Hansen N, Mac-Boima E, Rassin A, Betancourt TS. Alternate delivery platforms and implementation models for bringing evidence-based behavioral interventions to scale for youth facing adversity: a case study in West Africa. Implement Sci Commun. 2022 Feb 16;3(1):16. doi: 10.1186/s43058-022-00259-5. PMID 35168661
- [Derived] Betancourt TS, Hansen N, Farrar J, Borg RC, Callands T, Desrosiers A, Antonaccio CM, Williams MJ, Bangura J, Brennan RT. Youth Functioning and Organizational Success for West African Regional Development (Youth FORWARD): Study Protocol. Psychiatr Serv. 2021 May 1;72(5):563-570. doi: 10.1176/appi.ps.202000009. Epub 2020 Dec 9. PMID 33291974